CLINICAL TRIAL: NCT05667038
Title: Effect of Multi-Strain Probiotics as an Anti-Obesity Among Overweight and Obese Saudi Adults
Brief Title: Effect of Probiotics Among Overweight and Obese Saudi Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Hanan A Alfawaz, Prof, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-20-5503
Record Dates: First submitted 2022-12-07; First posted 2022-12-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Adult
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The study is a 12-week, a single center, double-blind, placebo-controlled, randomized, trial, 90 overweight or first-class obese subjects will be divided equally into two groups, a probiotics group, and a placebo group.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo arm (Placebo Comparator): The placebo sachets containing only the excipients, i.e., maize starch and maltodextrins, weights 3g. The placebo was indistinguishable in color, smell, and taste from the probiotic formulation.
  Interventions: Dietary Supplement: Placebo
- Probiotic arm (Experimental): Drug being used is Hexbio sachet containing 3g / 90 billion CFU. this drug is a formulation containing six microorganism strains (Lactobacillus acidophilus BCMC®12130, Lactobacillus casei subsp BCMC®12313, Lactobacillus lactis BCMC®12451, Bifidobacterium bifidum BCMC®02290, Bifidobacterium infantis BCMC®02129, and Bifidobacterium longum BCMC®02120).
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — The probiotics sachet contains a granular powder with 6 microorganism strains (30 × 109 CFU/gram): Lactobacillus acidophilus BCMC®12130, Lactobacillus casei subsp BCMC®12313, Lactobacillus lactis BCMC®12451, Bifidobacterium bifidum BCMC®02290, Bifidobacterium infantis BCMC®02129, and Bifidobacterium longum BCMC®02120.
  The drug is consumed orally, two sachets per day, by dissolving the sachet content in a glass of room-temperature water, one before breakfast and one before the last meal, for three months length.
  Other Names: (HEXBIO®) containing MCP® BCMC® strains
  Arms: Probiotic arm
Dietary Supplement: Placebo — Placebo:
  Subjects in the placebo group will receive the placebo consisting of only the carrier of the probiotic product, that is maize starch and maltodextrins.
  The sachet is consumed orally, two sachets per day, by dissolving the sachet content in a glass of room-temperature water, one before breakfast and one before the last meal, for three months length.
  Arms: Placebo arm

SUMMARY:
Obesity is classified as a low-grade chronic and systemic inflammatory disease and results from complicated interactions between genes and environmental factors, which leads to many diseases and affects the quality of life. There are growing interests in the effectiveness of probiotics as a supplementation to treat obesity through regulating microbiota host metabolism. Probiotics may influence the interplays among gut, brain, adipose, and liver in a way leading to weight. Since limited studies have been conducted on human subjects, more investigation is needed in this field. Therefore, this study sheds light on the investigation of the anti-obesity effect of probiotic supplementation.

DETAILED DESCRIPTION:
This study expects that the multi-strain probiotic product will induce beneficial changes in gut microbiota including reduction in weight, especially the visceral fat, which leads to reduction in systemic inflammatory state associated with fat accumulation. In order to evaluate the changes, ninety adult Saudi overweight or obese adult will be enrolled in this clinical trial and randomized to receive daily placebo or probiotics "MCP® BCMC® strains" for 12 weeks in a double-blind study. Biochemical markers will be measured through blood samples analyzed. Measurements and samples will be obtained at baseline and by the end of the study, at 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult's male and female ages between 19 to 40 years.
2. BMI (in kg/m2) from 25 to 35, (WHO, n. d.) Waist Circumference (WC) > 88 cm (women) or > 102 cm (men) (lean et al, 1995).
3. Stable body weight in the previous month of the trial.

Exclusion Criteria:

* Participants who suffer from diseases and on treatment, such as immune system diseases or thyroid disorders.
* Pregnant women or who plans to be pregnant.
* Participants who had gastrointestinal surgery.
* Hormone replacement therapy.
* Participants who taking antibiotic.
* Participants who consume probiotic or prebiotic supplementation regularly.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male & female
Enrollment: 90 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
waist circumference | 3 months
  The primary outcome in this study is the difference in waist circumference between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan A Alfawaz, Prof, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT05667038/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT05667038/ICF_001.pdf